CLINICAL TRIAL: NCT01026493
Title: A Randomized Phase I/II Study of ABT-888 in Combination With Temozolomide in Recurrent (Temozolomide Resistant) Glioblastoma
Brief Title: Veliparib and Temozolomide in Treating Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0929; CDR0000660545
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; recurrent adult brain tumor; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult brain stem glioma; adult mixed glioma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma | interventions — Temozolomide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase I: Dose Level 1 (Experimental): ABT-888 20 mg x 21 days plus temozolomide 60 mg x 21 days
  Interventions: Drug: temozolomide 60 mg x 21 days; Drug: ABT-888 20 mg x 21 days
- Phase I: Dose Level 2a (Experimental): ABT-888 40 mg x 21 days plus temozolomide 60 mg x 21 days
  Interventions: Drug: temozolomide 60 mg x 21 days; Drug: ABT-888 40 mg x 21 days
- Phase I: Dose Level 2b (Experimental): ABT-888 20 mg x 21 days plus temozolomide 75 mg x 21 days
  Interventions: Drug: temozolomide 75 mg x 21 days; Drug: ABT-888 20 mg x 21 days
- Phase I: Dose Level 3 (Experimental): ABT-888 40 mg x 21 days plus temozolomide 75 mg x 21 days
  Interventions: Drug: temozolomide 75 mg x 21 days; Drug: ABT-888 40 mg x 21 days
- Phase II: Arm 1/BEV-NAIVE (Experimental): ABT-888 40 mg x 21 days plus temozolomide 75 mg x 21 days
  Interventions: Drug: temozolomide 75 mg x 21 days; Drug: ABT-888 40 mg x 21 days
- Phase II: Arm 2/BEV-NAIVE (Experimental): ABT-888 40 mg x 5 days plus temozolomide 150 mg x 5 days
  Interventions: Drug: Temozolomide 150 mg x 5 days; Drug: ABT-888 40 mg x 5 days
- Phase II: Arm 1/BEV-FAILURE (Experimental): ABT-888 40 mg x 21 days plus temozolomide 75 mg x 21 days
  Interventions: Drug: temozolomide 75 mg x 21 days; Drug: ABT-888 40 mg x 21 days
- Phase II: Arm 2/BEV-FAILURE (Experimental): ABT-888 40 mg x 5 days plus temozolomide 150 mg x 5 days
  Interventions: Drug: Temozolomide 150 mg x 5 days; Drug: ABT-888 40 mg x 5 days

INTERVENTIONS:
Drug: temozolomide 60 mg x 21 days — Temozolomide 60 mg/m2 x 21 days, with a 28-day cycle. Treatment will continue until progressive disease unless toxicity or the discretion of the treating physician precludes further therapy.
  Other Names: Temodar; Temodal; Temcad
  Arms: Phase I: Dose Level 1; Phase I: Dose Level 2a
Drug: temozolomide 75 mg x 21 days — Temozolomide 75 mg/m2 x 21 days, with a 28-day cycle. Treatment will continue until progressive disease unless toxicity or the discretion of the treating physician precludes further therapy.
  Other Names: Temodar; Temodal; Temcad
  Arms: Phase I: Dose Level 2b; Phase I: Dose Level 3; Phase II: Arm 1/BEV-FAILURE; Phase II: Arm 1/BEV-NAIVE
Drug: ABT-888 20 mg x 21 days — 20 mg bid x 21 days, with a 28-day cycle. Treatment will continue until progressive disease unless toxicity or the discretion of the treating physician precludes further therapy.
  Other Names: Veliparib
  Arms: Phase I: Dose Level 1; Phase I: Dose Level 2b
Drug: ABT-888 40 mg x 21 days — 40 mg bid x 21 days/28-day cycle. Treatment continues until progressive disease unless toxicity or the discretion of the treating physician preclude further therapy
  Other Names: Veliparib
  Arms: Phase I: Dose Level 2a; Phase I: Dose Level 3; Phase II: Arm 1/BEV-FAILURE; Phase II: Arm 1/BEV-NAIVE
Drug: Temozolomide 150 mg x 5 days — 150 mg/m2 x 5 days (up to 200 mg/m2 after 2nd cycle)*, with a 28-day cycle; dose reduction to 125 mg/m2 if necessary. Treatment continues until progressive disease unless toxicity or the discretion of the treating physician preclude
  Other Names: Temodar; Temcad; Temodal
  Arms: Phase II: Arm 2/BEV-FAILURE; Phase II: Arm 2/BEV-NAIVE
Drug: ABT-888 40 mg x 5 days — 40 mg bid x 5 days/28-day cycle. Treatment continues until progressive disease unless toxicity or the discretion of the treating physician preclude
  Other Names: Veliparib
  Arms: Phase II: Arm 2/BEV-FAILURE; Phase II: Arm 2/BEV-NAIVE

SUMMARY:
RATIONALE: Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide. work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving veliparib together with temozolomide may kill more tumor cells.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of giving veliparib together with temozolomide and to see how well it works in treating patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define the maximum-tolerated dose of the combination of temozolomide and veliparib in patients with recurrent glioblastoma previously or not treated with temozolomide. (Phase I*)
* To determine the efficacy of the combination of temozolomide and veliparib (using a 5-day vs 21-day schedule) as measured by the 6-month progression-free survival rate in patients with recurrent glioblastoma previously treated with temozolomide. (Phase II*)

Secondary

* To characterize the safety profile of the combination of temozolomide and veliparib. (Phase I*)
* To determine the adverse event profile and tolerability of the combination of temozolomide and veliparib (using a 5-day vs 21-day schedule) in patients with recurrent glioblastoma. (Phase II*)
* To determine the efficacy of the combination of temozolomide and veliparib (using a 5-day vs 21-day schedule) as measured by objective response in patients with measurable disease. (Phase II*)
* To determine the overall survival of patients treated with the combination of temozolomide and veliparib (using a 5-day vs 21-day schedule). (Phase II*) Note: *Phase I was closed and phase II was opened on 3/6/12.

OUTLINE: This is a multicenter, phase I* dose-escalation study followed by a phase II* randomized study. Patients enrolled in the phase II portion are stratified according to bevacizumab (BEV) status (bevacizumab-naive vs bevacizumab-failure), age (< 50 years vs ≥ 50 years), Karnofsky performance status (70-80% vs 90-100%), and recent resection (yes vs no/biopsy only).

* Phase I:* Patients receive oral temozolomide once daily and oral veliparib twice daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Phase II:* Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive temozolomide and veliparib as in phase I.
  * Arm II: Patients receive oral temozolomide once daily and oral veliparib twice daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 1 year, every 26 weeks for 2 years, and then annually thereafter.

Note: *Phase I was closed and phase II was opened on 3/6/12.

PROJECTED ACCRUAL: A total of 240 patients (28 for phase I* and 212 for phase II*) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Any intracranial high-grade glioma (phase I*)
  * Glioblastoma or gliosarcoma (phase II*)
* Patients whose original histology was low-grade glioma are eligible provided they were subsequently diagnosed with glioblastoma or gliosarcoma
* Unequivocal radiographic evidence for tumor progression by MRI within 14 days prior to registration and with a stable or decreasing dose of steroids at least 5 days prior to scanning OR recent resection (registration within 30 days of resection) as long as all of the following conditions are met:

  * Patients must have recovered from the effects of surgery
  * Residual disease following resection of recurrent glioblastoma is not mandated for eligibility into the study; to best assess the extent of residual disease post-operatively, a post-operative MRI scan should be performed within 28 days prior to registration and within 96 hours post surgery (although 24 hours would be optimum)
  * Prior radiation is required for the phase I* arm
  * Patients must have completed a course of radiation therapy and at least 2 consecutive adjuvant cycles of temozolomide (phase II*)
  * A stable or decreasing dose of steroids at least 5 days prior to scanning is not mandated for patients who had a recent resection
* No evidence of acute (i.e., new and active) intratumoral hemorrhage on MRI

  * Patients with MRI demonstrating old hemorrhage or subacute blood after a neurosurgical procedure (biopsy or resection) are eligible Note: *Phase I was closed and phase II was opened on 3/6/12.

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* White blood cell (WBC) count ≥ 3,000/mm^3
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL (transfusion or other intervention allowed)
* Serum glutamic oxaloacetic transaminase (SGOT) ≤ 3.0 times upper limit of normal (ULN)
* Serum glutamic pyruvic transaminase (SGPT) ≤ 3.0 times ULN
* Bilirubin ≤ 1.25 times ULN
* Creatinine < 1.7 mg/dL OR estimated glomerular filtration rate (GFR) ≥ 30 mL/min
* Urine protein:creatinine ratio ≤ 0.5 OR urine protein < 1,000 mg by 24-hour urine collection**
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* Able to undergo brain MRI scans with IV gadolinium
* Able to swallow oral medications
* Patients with a history of seizure, or new onset of seizures, should be clinically controlled with no seizures for at least 14 days prior to registration
* No other prior invasive malignancy (except for nonmelanomatous skin cancer or carcinoma in situ of the cervix) unless the patient has been disease-free and off therapy for that disease for ≥ 3 years
* No severe, active comorbidity, including any of the following:

  * Transmural myocardial infarction or unstable angina within the past 6 months
  * Evidence of recent myocardial infarction or ischemia as indicated by S-T elevations of ≥ 2 mm on EKG performed within the past 14 days
  * New York Heart Association (NYHA) class II-IV congestive heart failure requiring hospitalization within the past 12 months
  * Stroke or transient ischemic attack within the past 6 months
  * Cerebral vascular accident within the past 6 months
  * Serious and inadequately controlled cardiac arrhythmia
  * Clinically significant peripheral vascular disease
  * Evidence of bleeding diathesis or coagulopathy
  * Serious non-healing would, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within the past 28 days
  * Significant traumatic injury within the past 28 days
  * Acute bacterial or fungal infection requiring IV antibiotics at the time of study registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within the past 14 days
  * AIDS based upon current Centers for Disease Control and Prevention (CDC) definition (HIV testing is not required)
* No condition that would impair the ability to swallow pills (e.g., GI tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease)
* No disease that would obscure toxicity or dangerously alter drug metabolism
* Not on dialysis
* No history of chronic hepatitis B or C Note: **Required for patients who received prior bevacizumab and developed known clinically significant nephrotic syndrome during treatment and whose baseline values have not returned to normal.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from the toxic effects of prior therapy
* Prior interstitial brachytherapy, Gliadel wafer, or stereotactic radiosurgery allowed provided there is confirmation of progressive disease by positron emission tomography (PET) scan, thallium scan, MRI spectroscopy, perfusion MRI, or surgical documentation
* No more than 3 prior treatment regimens (phase I*)
* No more than 2 prior treatment regimens for recurrent glioblastoma/gliosarcoma (phase II*)
* More than 28 days since prior major surgical procedure or open biopsy (with the exception of craniotomy)
* At least 28 days since prior investigational agents or cytotoxic agents (42 days for nitrosoureas, 21 days for procarbazine, and 14 days for vincristine)
* At least 14 days since prior non-cytotoxic agents (e.g., bevacizumab, interferon, tamoxifen, thalidomide, isotretinoin, or tyrosine kinase inhibitors)
* No concurrent highly-active antiretroviral therapy
* No concurrent herbal products of unknown constitution
* No concurrent major surgical procedures Note: *Phase I was closed and phase II was opened on 3/6/12.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Ian Robins, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Mark R Gilbert, MD, Principal Investigator — National Cancer Institute/National Institutes of Health; Arnab Chakravarti, MD, Study Chair — Arthur G. James Comprehensive Cancer Center and Richard J. Solove Research Institute, Ohio State University Medical School
Locations (17):
- United States (17):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - Leeward Radiation Oncology, ‘Ewa Beach, Hawaii
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Kansas City, Prairie Village, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II: Arm 1/BEV-NAIVE: ABT-888 40 mg x 5 days plus temozolomide 75 mg x 5 days
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2a | Phase I: Dose Level 2b | Phase I: Dose Level 3 | Phase II: Arm 1/BEV-NAIVE | Phase II: Arm 2/BEV-NAIVE | Phase II: Arm 1/BEV-FAILURE | Phase II: Arm 2/BEV-FAILURE
Started | 8 (Subjects with data available for the primary analysis are considered to have completed the study.) | 7 | 9 | 8 | 75 | 76 | 36 | 38
Completed | 8 | 6 | 9 | 8 | 73 | 73 | 32 | 37
Not Completed | 0 | 1 | 0 | 0 | 2 | 3 | 4 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 2 | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2a | Phase I: Dose Level 2b | Phase I: Dose Level 3 | Phase II: Arm 1/BEV-NAIVE | Phase II: Arm 2/BEV-NAIVE | Phase II: Arm 1/BEV-FAILURE | Phase II: Arm 2/BEV-FAILURE | Total
Number analyzed (Participants) | 8 | 6 | 9 | 8 | 73 | 73 | 32 | 37 | 246
Age, Continuous [Median (Full Range); unit: years] | 48 [20 to 63] | 51 [48 to 63] | 53 [18 to 67] | 41 [20 to 81] | 56 [21 to 77] | 56 [20 to 81] | 56 [20 to 70] | 57 [38 to 77] | 56 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 4 | 20 | 26 | 12 | 14 | 84
  Male | 6 | 5 | 4 | 4 | 53 | 47 | 20 | 23 | 162

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)
Description: Dose limiting toxicity (DLT) = any of the following events within 1st 8 weeks of treatment attributable to study drugs: Any grade (gr) 3/4 thrombocytopenia, gr 4 anemia, gr 3 neutropenia with fever (>100.4). gr 4 neutropenia lasting > 7 days; Any non-hematologic (NH) gr 3+ toxicity (TOX), excluding alopecia, despite maximal medical therapy (MLT); NH TOX such as rash, nausea, vomiting, diarrhea, mucositis, hypophosphatemia, and hypertension will only be considered DLTs if they remain gr 3+ despite MLT; 2nd occurrence of thromboembolism; Failure to recover from TOX (<= gr 1) to be eligible for re-treatment with study drugs <= 14 days of last dose of either drug; Any episode of non-infectious radiologically observed pneumonitis gr 2-4 any duration. Dose level will be considered acceptable if <= 1 of the 1st 6 eligible patients experiences a DLT. If current level is considered acceptable, dose escalation occurs. Otherwise preceding acceptable dose level will be declared the MTD.
Time Frame: Start of treatment to 8 weeks.
Population: Eligible patients who started study treatment
Measure: Number; unit: participants
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2a | Phase I: Dose Level 2b | Phase I: Dose Level 3
Number analyzed (Participants) | 8 | 6 | 9 | 8
participants | 1 | 0 | 1 | 1

2. Primary Outcome: Phase II: 6-month Progression-free Survival (PFS) Rate for Patients With Measurable Disease After Surgery
Description: For patients with measureable disease after surgery: Progression defined as ≥ 25% increase in size of enhancing tumor or any new tumor; or neurologically worse, and steroids stable/increased. Bevacizumab (BEV)-naïve group: p0= 15% as estimate of 6-mo. PFS [null hypothesis (NH)], p1= 30%, with a 15% absolute increase [alternative hypothesis (AH)]. Error rates of 10% alpha and 10% beta. If <= 11 patients experience 6-month PFS of the first 53 analyzable patients, then do not reject the null hypothesis that the 6-month PFS rate of experimental arm is less than 15%; BEV-failure group: p0 = 2% as a conservative estimate of 6-month PFS [NH], p1 = 15%, with a 13% absolute increase [AH]. Using first 26 analyzable subjects for each experimental arm, there is >= 90% power to detect >= 15% increase at a significance level of 0.10, using a 1-sided binomial test. If >= 2 patients (8%) are progression free at 6 mo., then claim this regimen to be promising in the patient group.
Time Frame: Randomization to 6 months.
Population: Randomized patients with measurable disease after surgery, at least one cycle of treatment, evaluable for 6 month PFS, and within the required sample size (i.e. the first 53 BEV-naive patients and the first 26 BEV-failure patients- the number of patients will be less than sample size if not enough patients meet the criteria).
Measure: Number; unit: participants
Arm/Group | Phase II: Arm 1/BEV-NAIVE | Phase II: Arm 2/BEV-NAIVE | Phase II: Arm 1/BEV-FAILURE | Phase II: Arm 2/BEV-FAILURE
Number analyzed (Participants) | 53 | 53 | 19 | 26
participants | 9 | 9 | 1 | 1

3. Secondary Outcome: Phase II: Objective Response (Partial and Complete Response) Rate for Patients With Measurable Disease After Surgery
Description: Response and progression will be evaluated using standard criteria for patients with malignant gliomas (Macdonald 1990). Partial response and complete response are centrally reviewed.
Time Frame: Analysis occurs after all patients have been on study for at 6 months. (Patients are followed from randomization to death or study termination whichever occurs first.)
Population: Eligible patients with at least one cycle of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Arm 1/BEV-NAIVE | Phase II: Arm 2/BEV-NAIVE | Phase II: Arm 1/BEV-FAILURE | Phase II: Arm 2/BEV-FAILURE
Number analyzed (Participants) | 53 | 53 | 19 | 26
percentage of participants | 0 [0 to 0] | 3.8 [0 to 8.9] | 5.3 [0 to 15.3] | 0 [0 to 0]

4. Secondary Outcome: Phase II: Overall Survival (OS)
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. This analysis was planned to occur when all patients had been potentially followed for at least 6 months.
Time Frame: as for outcome 3
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm 1/BEV-NAIVE | Phase II: Arm 2/BEV-NAIVE | Phase II: Arm 1/BEV-FAILURE | Phase II: Arm 2/BEV-FAILURE
Number analyzed (Participants) | 73 | 73 | 32 | 37
months | 10.3 [7.6 to 13.4] | 10.7 [7.6 to 12.6] | 4.7 [3.0 to 6.3] | 4.7 [3.4 to 7.0]
Statistical Analysis 1: Comparison: Phase II: Arm 1/BEV-NAIVE vs Phase II: Arm 2/BEV-NAIVE; Test type: Superiority or Other; p = 0.95, Log Rank; Two-sided test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.66 to 1.48] — Reference level = Arm 1/BEV-NAIVE
Statistical Analysis 2: Comparison: Phase II: Arm 1/BEV-FAILURE vs Phase II: Arm 2/BEV-FAILURE; Test type: Superiority or Other; p = 0.93, Log Rank; Two-sided test; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.57 to 1.53] — Reference level = Arm 1/BEV-FAILURE

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2a | Phase I: Dose Level 2b | Phase I: Dose Level 3 | Phase II: Arm 1/BEV-NAIVE | Phase II: Arm 2/BEV-NAIVE | Phase II: Arm 1/BEV-FAILURE | Phase II: Arm 2/BEV-FAILURE
Serious Adverse Events (participants affected / at risk) | 2/8 | 2/6 | 1/9 | 6/8 | 19/73 | 15/73 | 14/32 | 10/37
Other Adverse Events (participants affected / at risk) | 7/8 | 5/6 | 9/9 | 6/8 | 70/73 | 70/73 | 31/32 | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1 (N=8) | Phase I: Dose Level 2a (N=6) | Phase I: Dose Level 2b (N=9) | Phase I: Dose Level 3 (N=8) | Phase II: Arm 1/BEV-NAIVE (N=73) | Phase II: Arm 2/BEV-NAIVE (N=73) | Phase II: Arm 1/BEV-FAILURE (N=32) | Phase II: Arm 2/BEV-FAILURE (N=37)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Death NOS (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 5 | 0 | 1 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 3 | 0 | 5 | 1
White blood cell decreased (Investigations) | 0 | 0 | 0 | 2 | 3 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 3 | 1 | 6 | 4
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Edema cerebral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1 | 5 | 4 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1 (N=8) | Phase I: Dose Level 2a (N=6) | Phase I: Dose Level 2b (N=9) | Phase I: Dose Level 3 (N=8) | Phase II: Arm 1/BEV-NAIVE (N=73) | Phase II: Arm 2/BEV-NAIVE (N=73) | Phase II: Arm 1/BEV-FAILURE (N=32) | Phase II: Arm 2/BEV-FAILURE (N=37)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 3 | 24 | 25 | 8 | 11
Vitreous hemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 4 | 1 | 20 | 12 | 11 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 3 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 19 | 23 | 8 | 3
Edema limbs (General disorders) | 1 | 1 | 0 | 1 | 4 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 2 | 5 | 4 | 36 | 36 | 16 | 18
Pain (General disorders) | 1 | 0 | 0 | 1 | 2 | 4 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3 | 4 | 10 | 16 | 6 | 3
Lymphocyte count decreased (Investigations) | 1 | 1 | 6 | 3 | 31 | 31 | 12 | 13
Neutrophil count decreased (Investigations) | 1 | 0 | 2 | 2 | 25 | 15 | 7 | 3
Platelet count decreased (Investigations) | 1 | 1 | 6 | 3 | 39 | 48 | 16 | 22
White blood cell decreased (Investigations) | 1 | 1 | 4 | 5 | 32 | 28 | 11 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3 | 17 | 18 | 9 | 10
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 4 | 7 | 3 | 4
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 4 | 3 | 4 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 5 | 3
Cognitive disturbance (Nervous system disorders) | 2 | 0 | 0 | 1 | 6 | 5 | 2 | 2
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 1 | 5 | 4 | 2 | 3
Headache (Nervous system disorders) | 2 | 1 | 5 | 2 | 28 | 26 | 10 | 8
Hypersomnia (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 1 | 4 | 0 | 5 | 12 | 3 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Seizure (Nervous system disorders) | 2 | 1 | 0 | 1 | 14 | 10 | 4 | 4
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 7 | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 4 | 5 | 3 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 2 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 6 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 2 | 1 | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.